CLINICAL TRIAL: NCT02059187
Title: A Phase III Clinical Trial to Study the Safety and Efficacy of MK-1293 Compared to Lantus™ in Subjects With Type 2 Diabetes Mellitus
Brief Title: The Safety and Efficacy of MK-1293 Versus Lantus™ in Participants With Type 2 Diabetes Mellitus (MK-1293-006)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1293-006; 2012-003478-19 (EudraCT Number)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — MK-1293; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-1293 (Experimental): MK-1293 administered subcutaneously once daily in the evening.
  Interventions: Drug: MK-1293; Drug: Prandial insulin
- Lantus™ (Active Comparator): Lantus™ administered subcutaneously once daily in the evening.
  Interventions: Drug: Lantus™; Drug: Prandial insulin

INTERVENTIONS:
Drug: MK-1293 — MK-1293 (insulin glargine) 100 units/mL administered subcutaneously once daily for 24 weeks. Participants not taking insulin at study entry will initiate MK-1293 at 10 units daily. Participants taking insulin will initiate MK-1293 at an appropriate dose based on prior insulin dosing. After initiation, the dose will be titrated to the suggested target for fasting finger stick glucose. MK-1293 dosing once daily at times other than bedtime will be permitted for participants with a previously established dosing time.
  Arms: MK-1293
Drug: Lantus™ — Lantus™ (insulin glargine [rDNA origin]) 100 units/mL administered subcutaneously once daily for 24 weeks. Participants not taking insulin at study entry will initiate Lantus™ at 10 units daily. Participants taking insulin will initiate Lantus™ at an appropriate dose based on prior insulin dosing. After initiation, the dose will be titrated to the suggested target for fasting finger stick glucose. Lantus™ dosing once daily at times other than bedtime will be permitted for participants with a previously established dosing time.
  Other Names: Insulin glargine [rDNA origin]
  Arms: Lantus™
Drug: Prandial insulin — Participants taking prandial insulin will continue their current prandial insulin regimen during the insulin glargine titration. After the insulin glargine titration phase, the prandial insulin may be adjusted if the investigator determines it to be necessary for glucose control.

SUMMARY:
This 24-week study is a safety and efficacy comparison of MK-1293 and Lantus™ in participants with type 2 diabetes mellitus (T2DM). The primary hypothesis is that after 24 weeks, the mean change in hemoglobin A1c (A1C) from baseline is non-inferior (with margin of 0.4%) in participants treated with MK-1293 compared with that in participants treated with Lantus™.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes Mellitus (T2DM) as defined by the American Diabetes Association (ADA) or the European Association for the Study of Diabetes (EASD)
* hemoglobin A1C of ≤11.0% and requires insulin for glycemic control
* Body mass index (BMI) <45 kg/m^2

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis, or has type 1 diabetes confirmed with a C-peptide <0.7 ng/mL (0.23 nmol/L)
* One or more severe hypoglycemic episodes associated with hypoglycemic seizures, comas or unconsciousness within the past 6 months
* History of intolerance or hypersensitivity to Lantus™ or contraindication to Lantus™ or one of its excipients based on the label of the country of the investigational site
* On a weight loss program within the last 8 weeks
* Received injectable incretin-based therapy (e.g., Victoza™, Byetta™) within the prior 8 weeks
* Bariatric surgery within 12 months prior to signing the informed consent
* Likely to require treatment for ≥2 consecutive weeks or repeated courses of corticosteroids
* Undergone a surgical procedure within 4 weeks prior to signing informed consent or has planned major surgery during the study
* New or worsening signs or symptoms of coronary heart disease or congestive heart failure within the last 3 months
* Presence of any of the following during the last 3 months: acute coronary syndrome, coronary artery intervention, and/or stroke or transient ischemic neurological disorder
* Severe peripheral vascular disease
* Systolic blood pressure ≥ 160 mm Hg or a diastolic ≥95 mm Hg and blood pressure is not considered likely to be under these limits with an adjustment in antihypertensive medication
* Chronic myopathy or a progressive neurological or neuromuscular disorder
* Active nephropathy
* History of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
* Human immunodeficiency virus (HIV)
* Clinically important hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* History of malignancy ≤5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* History of melanoma, leukemia, lymphoma, or renal cell carcinoma
* Hyperthyroidism
* On a stable dose of thyroid hormone replacement therapy for <6 weeks
* Uses recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence
* Pregnant or breast-feeding, or is expecting to conceive or donate eggs during the study, including 14 days following the last dose of study drug
* Donated blood products or has had phlebotomy of >300 mL within 8 weeks of signing informed consent, or intends to donate blood products within the projected duration of the study
* Poor mental function or any other reason to expect that the participant may have difficulty in complying with the requirements of the study
* Clinically significant ECG abnormality which exposes the participant to risk by enrolling in the study
* Positive urine pregnancy test
* Participant is a night shift worker which causes difficulty complying with the overnight fast requirement and has potential for confounding the 7-point SMBG analysis
* Participant, as assessed by the investigator, is not appropriate for or does not agree to target a fasting glucose of 70-100 mg/dL [3.9 -5.6 mmol/L]
* Has used a formulation of glargine insulin other than Lantus™

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2014-02-11 (Actual); Primary Completion 2015-03-11 (Actual); Study Completion 2015-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Hollander PA, Carofano WL, Lam RLH, Golm GT, Eldor R, Crutchlow MF, Marcos MC, Rendell MS, Home PD, Gallwitz B, Rosenstock J. Efficacy and safety of MK-1293 insulin glargine compared with originator insulin glargine (Lantus) in type 2 diabetes: A randomized, open-label clinical trial. Diabetes Obes Metab. 2018 Sep;20(9):2229-2237. doi: 10.1111/dom.13363. Epub 2018 Jun 10. PMID 29761615

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-1293: MK-1293 administered subcutaneously once daily.
- Lantus™: Lantus™ administered subcutaneously once daily.
Period: Overall Study
Arm/Group | MK-1293 | Lantus™
Started | 265 | 266
Completed | 240 | 244
Not Completed | 25 | 22
Not completed — Adverse Event | 0 | 3
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 9 | 8
Not completed — Non-compliance with study drug | 1 | 0
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 12 | 8

BASELINE CHARACTERISTICS:
Population: The analysis population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1293 | Lantus™ | Total
Number analyzed (Participants) | 265 | 266 | 531
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.9 (10.0) [20 to 80] | 57.1 (9.8) [31 to 79] | 57.0 (9.9) [20 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 125 | 238
  Male | 152 | 141 | 293

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Participant Hemoglobin A1C Level at Week 24
Description: A1C is measured as a percent. A1C is the key glycemic parameter which correlates with reduction of risk of diabetic complications.
Time Frame: Baseline and Week 24
Population: The analysis population included all randomized, treated participants who had at least one observation for the analysis endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent A1C
Arm/Group | MK-1293 | Lantus™
Number analyzed (Participants) | 263 | 263
Percent A1C | -1.28 [-1.41 to -1.15] | -1.30 [-1.43 to -1.18]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus™; Test type: Non-Inferiority or Equivalence — MK-1293 was to be considered non-inferior to Lantus in type 2 diabetes mellitus (T2DM) if the upper bound of the two-sided 95% confidence interval (CI) for the between-treatment difference (MK-1293 minus Lantus) in least-squares (LS) means was below 0.4% based on a cLDA model; Difference in least squares means = 0.03, 95% CI 2-sided [-0.12 to 0.18]

2. Primary Outcome: Percentage of Participants With Confirmed Anti-Insulin Antibodies (AIA) up to Week 24
Description: Percentage of participants is a cumulative percentage of participants with any confirmed AIA (including baseline) up to Week 24.
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1293 | Lantus™
Number analyzed (Participants) | 262 | 262
Percentage of participants | 34.7 | 29.0
Statistical Analysis 1: Comparison: MK-1293 vs Lantus™; Test type: Superiority or Other; Difference in percentage = 5.7, 95% CI 2-sided [-2.3 to 13.7]

3. Secondary Outcome: Change From Baseline in Participant Body Weight at Week 24
Description: Change from baseline in participant body weight at Week 24.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | MK-1293 | Lantus™
Number analyzed (Participants) | 242 | 246
kilograms | 1.3 (3.6) | 1.4 (4.5)

4. Secondary Outcome: Percentage of Participants Experiencing an Adverse Event (AE) of Hypoglycemia Up to Week 24
Description: Symptomatic events assessed as likely to be hypoglycemia were to be reported by investigators as adverse events of hypoglycemia; a concurrent glucose measurement was not required. Asymptomatic events with confirmed glucose levels </= 70mg/dL (</= 3.9mmol/L) could also be reported as adverse events at the discretion of the investigator.
Time Frame: Up to 24 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1293 | Lantus™
Number analyzed (Participants) | 263 | 263
Percentage of participants | 54.0 | 54.0
Statistical Analysis 1: Comparison: MK-1293 vs Lantus™; Test type: Superiority or Other; Difference in percentage = 0.0, 95% CI 2-sided [-8.5 to 8.5]

5. Secondary Outcome: Percentage of Participants Experiencing an AE Over the 24-week Treatment Period
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the investigational product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the investigational product, is also an AE.
Time Frame: Up to 24 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1293 | Lantus™
Number analyzed (Participants) | 263 | 263
Percentage of participants | 78.3 | 71.5
Statistical Analysis 1: Comparison: MK-1293 vs Lantus™; Test type: Superiority or Other; Difference in percent = 6.8, 95% CI 2-sided [-0.6 to 14.2]

6. Secondary Outcome: Daily Basal Insulin Dose (Units) at Week 24
Description: The daily basal insulin dose (measured in units) for any given visit is defined as the average dose from the three most recent days preceding the visit date.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units
Arm/Group | MK-1293 | Lantus™
Number analyzed (Participants) | 263 | 262
Units | 48.2 [44.9 to 51.5] | 46.9 [43.5 to 50.2]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus™; Test type: Superiority or Other; Difference in LS means = 1.4, 95% CI 2-sided [-2.2 to 4.9]

7. Secondary Outcome: Daily Basal Insulin Dose Per Body Weight (Units/kg) at Week 24
Description: Basal insulin dose per body weight was calculated as total insulin dose (units) per day divided by body weight in kilograms (kg).
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units/kg
Arm/Group | MK-1293 | Lantus™
Number analyzed (Participants) | 263 | 262
Units/kg | 0.53 [0.49 to 0.56] | 0.51 [0.48 to 0.54]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus™; Test type: Superiority or Other; Dofference in LS means = 0.01, 95% CI 2-sided [-0.02 to 0.05]

8. Secondary Outcome: Change From Baseline in Participant Fasting Plasma Glucose (FPG) at Week 24
Description: Participants fasted (no food or drink except water and non-antihyperglycemic non-study medications as prescribed) for at least 8 hours prior to all study visits.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-1293 | Lantus™
Number analyzed (Participants) | 263 | 263
mg/dL | -35.0 [-41.3 to -28.6] | -38.4 [-44.8 to -32.1]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus™; Test type: Superiority or Other; Difference in LS means = 3.5, 95% CI 2-sided [-3.7 to 10.7]

9. Secondary Outcome: Change From Baseline in Participant 7-Point Average of Self-Monitored Blood Glucose (SMBG) at Week 24
Description: 7-Point Average of SMBG was defined as the mean of blood glucose measurements taken at the following 7 times: before morning meal, after morning meal, before midday meal, after midday meal, before evening meal, after evening meal or at bedtime, and between 2 AM and 4 AM.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-1293 | Lantus™
Number analyzed (Participants) | 246 | 235
mg/dL | -30.7 [-37.6 to -23.8] | -27.3 [-34.0 to -20.5]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus™; Test type: Superiority or Other; Difference in LS Means = -3.4, 95% CI 2-sided [-11.3 to 4.4]

10. Secondary Outcome: Percentage of Participants With Hemoglobin A1C <7% at Week 24
Description: Percentage of participants with A1C <7.0% (53 mmol/mol) at Week 24.
Time Frame: Week 24
Population: The analysis population included all randomized, treated participants with a Week 24 A1C measurement.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1293 | Lantus™
Number analyzed (Participants) | 241 | 245
Percentage of participants | 46.5 | 43.7
Statistical Analysis 1: Comparison: MK-1293 vs Lantus™; Test type: Superiority or Other; Adjusted difference in percent = 2.8, 95% CI 2-sided [-6.1 to 11.6] — Calculated via Miettinen and Nurminen method, stratified by prior insulin status

11. Secondary Outcome: Percentage of Participants With Hemoglobin A1C <6.5% at Week 24
Description: Percentage of participants with A1C <6.5% (48 mmol/mol) at Week 24.
Time Frame: Week 24
Population: The analysis population included all randomized, treated participants with a Week 24 A1C measurement.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1293 | Lantus™
Number analyzed (Participants) | 241 | 245
Percentage of participants | 21.6 | 22.4
Statistical Analysis 1: Comparison: MK-1293 vs Lantus™; Test type: Superiority or Other; Adjusted difference in percent = -0.9, 95% CI 2-sided [-8.3 to 6.5] — Calculated via Miettinen and Nurminen method, stratified by prior insulin status

ADVERSE EVENTS:
Time Frame: Up to 26 weeks (including 2-week follow-up for serious adverse events)
Description: All randomized participants who received at least one dose of study treatment.
Arm/Group | MK-1293 | Lantus™
Serious Adverse Events (participants affected / at risk) | 13/263 | 9/263
Other Adverse Events (participants affected / at risk) | 147/263 | 151/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1293 (N=263) | Lantus™ (N=263)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve disease mixed (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1293 (N=263) | Lantus™ (N=263)
Upper respiratory tract infection (Infections and infestations) | 16 (16) | 15 (16)
Hypoglycaemia (Metabolism and nutrition disorders) | 142 (1352) | 142 (1141)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.